CLINICAL TRIAL: NCT05414994
Title: Assessment of the Ocular Microbiome in Health and Disease
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sapna Gangaputra, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 10001
Record Dates: First submitted 2022-05-19; First posted 2022-06-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Microbial Colonization; Eye Diseases; Ophthalmopathy
MeSH Terms: conditions — Communicable Diseases; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The inner eyelid of both eyelids will be swabbed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort A: normal eyes with no ocular disease
  Interventions: Other: Eye swab
- Cohort B: primary open angle glaucoma/Ocular hypertension defined as mild glaucoma which is well controlled with no more than one drop of prostaglandin use daily for the past 6 months
  Interventions: Other: Eye swab
- Cohort C: non-infectious keratopathy not using any prescription medication (OTC artificial tears are acceptable)
  Interventions: Other: Eye swab
- Cohort D: Dry AMD (age related macular degeneration)
  Interventions: Other: Eye swab
- Cohort E: Wet AMD
  Interventions: Other: Eye swab
- Cohort F: diabetic retinopathy, any stage
  Interventions: Other: Eye swab

INTERVENTIONS:
Other: Eye swab — This is a simple swab under the eyelids of both eyes

SUMMARY:
The objective of this application is to illustrate the core constituents of the ocular surface microbiome, describe factors that promote colonization, and assess the ocular microbiome's role in the health of the anterior segment. We will conduct a prospective, observational cohort study, including a longitudinal analysis of the ocular microbiome in adults.

DETAILED DESCRIPTION:
The microbiome is defined as a community of microbial organisms that reside in a specific host niche. There is a growing body of literature on the association between gut microbiome and disease entities such as inflammatory bowel disease, colon cancer and presumably an association that might influence response to treatment in some patients.

Recent data suggest the existence of a resident ocular microbiota that may play a protective role in corneal infections [1-4]. However, not much is known about the ocular microbiome and its association with disease or response to treatment. The National Eye Institute (NEI) recently hosted a symposium to discuss challenges to characterize the ocular microbiome and its role in promoting or preventing ocular diseases. One of the major challenges discussed is the lack of a normative population- based database describing the ocular microbiome.

In response the NEI as part of the Anterior segment initiative put out an RFA requesting proposals on methods of collection of biological samples and associated clinical data (e.g. demographic, residence, medications, allergies); processing of samples to extract analytes (e.g., DNA, RNA, protein, metabolites) and characterizing microorganisms in a low biomass niche, specifically the ocular surface using16S rRNA marker gene, whole metagenome sequencing (WMS), and metatranscriptomics approaches.

ELIGIBILITY:
Inclusion Criteria:

We will include subjects who meet all of the following criteria:

* 18 years of age or older
* Provide informed consent
* Cohort A - normal eyes with no ocular disease
* Cohort B - primary open angle glaucoma/Ocular hypertension defined as mild glaucoma which is well controlled with no more than one drop of prostaglandin use daily for the past 6 months
* Cohort C - non-infectious keratopathy not using any prescription medication (OTC artificial tears are acceptable)
* Cohort D - Dry AMD (age related macular degeneration)
* Cohort E - Wet AMD
* Cohort F - diabetic retinopathy

Exclusion Criteria:

We will exclude subjects who meet all of the following criteria:

* Prior ocular disease either of the anterior or posterior segment
* Any medical comorbidities except well controlled DH and HTN
* Unable to follow up with study procedures as described

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We anticipate there will be approximately 20% failure rate due to the low bacterial load in these samples and so we will have to collect more samples to account for the loss of data.
  We estimate that 20 patients in each cohort of eyes with ocular disease - 100 total patients and 500 normal eyes will give us sufficient power to explore this topic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Normal Ocular Microbiome | 3 years
  Number of patients in middle Tennessee with a normal ocular microbiome by development of a normative database.

SECONDARY OUTCOMES:
Whole Metagenome Sequencing Methods | 3 years
  Number of ocular microbial species in different age and ethnic groups by the development of whole metagenome sequencing methods optimized for low biomass samples to characterize the ocular surface (anterior segment) microbiome.

OTHER OUTCOMES:
Novel Metatranscriptomics Analysis | 3 years
  Number of active microbial pathways and host epithelial gene expression profiles by novel metatranscriptomics analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No